CLINICAL TRIAL: NCT02626312
Title: Phase I Trial of Radiation Therapy in Patients With Liver Cancers and Impaired Liver Function
Brief Title: Radiation Therapy in Treating Patients With Hepatocellular Carcinoma, Cholangiocarcinoma, or Liver Metastasis Who Have Impaired Liver Function
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0052; P30CA016672 (NIH); NCI-2016-00006 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0052 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cholangiocarcinoma; Cirrhosis; Hepatocellular Carcinoma; Metastatic Malignant Neoplasm in the Liver
MeSH Terms: conditions — Cholangiocarcinoma; Fibrosis; Carcinoma, Hepatocellular | interventions — Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy) (Experimental): Patients undergo radiation therapy 5 days a week for a total of 15 or 25 fractions in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Other: Survey Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Correlative studies
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and the best dose of radiation therapy in treating patients with hepatocellular carcinoma, cholangiocarcinoma, or cancer that has spread from the original (primary) tumor to the liver who also have impaired liver function (liver damage caused by cirrhosis, chemotherapy, or surgery). Radiation therapy (RT) uses high energy x-rays to kill tumor cells and shrink tumors. New methods of giving RT to the liver may help control cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of high dose radiotherapy in patients who have liver tumors (hepatocellular carcinoma [HCC]/cholangiocarcinoma/liver metastases from any primary) and who have impaired liver function or low functional liver volume or who have received prior liver radiation.

SECONDARY OBJECTIVES:

I. To evaluate 2 year local control with radiotherapy in these patients. II. To evaluate tumor response, patterns of failure, and survival in these patients.

III. To evaluate imaging- and serum-based biomarkers in these patients, as correlates of hepatic toxicity and tumor response.

OUTLINE: This is a dose-escalation study.

Patients undergo radiation therapy 5 days a week for a total of 15 or 25 fractions in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4-8 weeks and then every 3-4 months for 2 years. Patients who progress during the two year follow-up period are followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma, cholangiocarcinoma, or liver metastasis from any histology
* Patients may have single or multinodular tumors
* There is no specific tumor size cut-off for this protocol; however, the radiation treatment plan must meet the protocol's dose constraints
* Compromised liver function as defined by any of the following:

  * Cohort 1: Advanced cirrhosis group

    * Borderline Child-Pugh class A6
    * Child-Pugh class B

      * The patients in this advanced cirrhosis group must have at least 400 ml of functional liver, as estimated on either diagnostic imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) or single photon emission computed tomography (SPECT)/CT with Tc-99m sulfur colloid; there is no upper limit on the functional liver volume for these patients
  * Cohort 2: Low functional liver volume without underlying chronic liver disease

    * Previous irinotecan or oxaliplatin chemotherapy
    * Previous liver resection(s)

      * These patients must have at least 400 ml of functional liver, as estimated by either diagnostic imaging computed tomography or magnetic resonance imaging (CT or MRI) or SPECT/CT with Tc-99m sulfur colloid; there is no upper limit on the functional liver volume for these patients;
  * Cohort 3: History of prior liver-directed radiation therapy with either fractionated external beam radiation therapy (EBRT), stereotactic body radiation therapy (SBRT) or yttrium-90 radioembolization (Y90 RE); the interval between prior EBRT and re-irradiation on protocol should be equal to or greater than 12 months; the interval between prior Y90 RE and re-irradiation on protocol should be equal to or greater than 6 months;

    * Cirrhosis group:

      * Child-Pugh class A5;
      * Borderline Child-Pugh class A6;
      * The patients in this group must have at least 400 ml of functional liver, as estimated on either diagnostic imaging (CT or MRI) or SPECT/CT with Tc-99m sulfur colloid; there is no upper limit on the functional liver volume for these patients
  * Low functional liver volume without underlying liver disease

    * Previous irinotecan or oxaliplatin chemotherapy
    * Previous liver resection(s)
    * These patients must have at least 400 ml of functional liver, as estimated by either diagnostic imaging (CT or MRI) or SPECT/CT with Tc-99m sulfur colloid; there is no upper limit on the functional liver volume for these patients
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Women of childbearing potential (those who have not undergone a hysterectomy or who have not been postmenopausal for at least 24 consecutive months) must agree to practice adequate contraception and to refrain from breast feeding
* Prior history of surgical resection, chemotherapy, transarterial chemoembolization (TACE), and/or radiofrequency ablation are allowed
* Expected survival must be greater than 3 months
* Patients may receive concurrent capecitabine or sorafenib at the discretion of the treating physicians
* Signed study-specific consent form

Exclusion Criteria:

* Prior liver-directed radiation therapy in cohort 1 (advanced cirrhosis group) or cohort 2 (low functional volume group)
* Prior yttrium-90 therapy for patients in cohorts 1 or 2
* Patients with a Child-Pugh score less than 6 or greater than 9 for radiation naive patients with cirrhosis (cohort 1)
* Child-Pugh score of greater than 6 for patients with cirrhosis who previously received liver directed radiation (EBRT or Y90 RE) (cohort 3)
* Unstable angina and/or symptomatic congestive heart failure requiring hospitalization within the last 6 months; transmural myocardial infarction within the last 6 months prior to study entry
* Current evidence of fever or untreated infection
* Active hepatitis, including but not limited to viral and drug-induced
* Poorly controlled inflammatory bowel disease
* Women with a positive pregnancy test
* Inability to comply with study and/or follow-up procedures
* Patients with an active second malignancy or prior invasive malignancy unless disease free for a minimum of 3 years; non-melanoma skin cancer and previous early prostate cancer that had a non-rising prostate-specific antigen (PSA) can be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Maximum dose constraint | 4-8 weeks after completion of radiation therapy
  Defined as the highest level dose constraint at which no more than 1 of 6 evaluable patients has had a dose limiting toxicity. Toxicities will be summarized with frequency by type, severity and their relationship to the treatment.

SECONDARY OUTCOMES:
Local disease control rate | Up to 2 years
  The Kaplan Meier method will be used to estimate 2-year local disease control rate.
Tumor response | Up to 2 years
  Will be observed.
Patterns of failure | Up to 2 years
  Will be observed.
Overall survival | Up to 2 years
  The Kaplan Meier method will be used to estimate the probability of overall survival.

OTHER OUTCOMES:
Tumor biomarker expression in serum | Baseline
  Imaging- and serum-based biomarkers will be correlated with hepatic toxicity and tumor response. Plots such as box plot and scatter plots will be used to evaluate expressions of markers between patients with and without response, and between patients having experienced DLTs and patients having not experienced DLTs, and Wilcoxon rank sum test will be used to compare expressions of markers between these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J Koay, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chang E, Wong FCL, Chasen BA, Erwin WD, Das P, Holliday EB, Koong AC, Ludmir EB, Minsky BD, Noticewala SS, Smith GL, Taniguchi CM, Rodriguez MJ, Beddar S, Martin-Paulpeter RM, Niedzielski JS, Sawakuchi GO, Schueler E, Perles LA, Xiao L, Szklaruk J, Park PC, Dasari AN, Kaseb AO, Kee BK, Lee SS, Overman MJ, Willis JA, Wolff RA, Tzeng CD, Vauthey JN, Koay EJ. Phase I trial of single-photon emission computed tomography-guided liver-directed radiotherapy for patients with low functional liver volume. JNCI Cancer Spectr. 2024 Apr 30;8(3):pkae037. doi: 10.1093/jncics/pkae037. PMID 38730548